CLINICAL TRIAL: NCT02217189
Title: Study of the Effect of Oral Zinc Supplementation on Superoxide Radical Scavengers in Spermatozoa of Patients With Asthenospermia
Brief Title: Study of the Effect of Oral Zinc Supplementation on Superoxide Radical Scavengers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Babylon University (Other)
Collaborators: Ministry of Health, Iraq (Network)
Responsible Party: Principal Investigator, mahmoud hussein hadwan, Mahmoud Hussein Hadwan, Babylon University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Babil-3
Record Dates: First submitted 2014-08-06; First posted 2014-08-15 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Asthenozoospermia
Keywords: Zinc supplementation.; Oxidative stress.; Superoxide radical scavengers.; Asthenospermia.; Oxido-sensitive index.
MeSH Terms: conditions — Asthenozoospermia | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc sulfate (Experimental): 60 subfertile (age 32.5±3.23 year) men with asthenozoospermia was treated with zinc sulfate, every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Interventions: Dietary Supplement: zinc sulfate
- Healthy control (No Intervention): 60 fertile (age 31.6±3.3 year) men, no treatment.

INTERVENTIONS:
Dietary Supplement: zinc sulfate — The subfertile group treated with zinc sulfate, every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Arms: Zinc sulfate

SUMMARY:
Although several studies have considered the relationship between infertility and semen super oxide radical scavengers levels, no study on the effects of asthenospermia treatments such as oral zinc supplementation on superoxide radical scavengers activity which are important in fertility of the individual has been reported.

DETAILED DESCRIPTION:
The present study was conducted to study the effect of zinc supplementation on the quantitative and qualitative characteristics of semen along with superoxide radical scavengers activity in the seminal plasma of asthenospermic patients.

ELIGIBILITY:
Inclusion Criteria:

* the presence of asthenozoospermia in the semen sample.

Exclusion Criteria:

* the absence of endocrinopathy, varicocele, and female factor infertility. Smokers and alcoholic men were excluded from the study because of their recognized high seminal ROS levels and decreased antioxidant levels.

Ages: 26 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Oxido-sensitive index level in spermatozoa and seminal plasma. | up to three months.

SECONDARY OUTCOMES:
Volume of semen. | up to three months.
Xanthine oxidase activity in spermatozoa and seminal plasma. | up to three months.
Catalase like activity in spermatozoa and seminal plasma. | up to three months.
Superoxide dismutase activity in spermatozoa and seminal plasma. | up to three months.
Progressive sperm motility percentage. | up to three months
Total normal sperm count. | up to three months.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud H. Hadwan, PhD, Principal Investigator — Babylon University/ Iraq; Lamia A. Almashhedy, PhD, Study Director — Babylon University/ Iraq; Abdulrrazaq S. Alsalman, PhD, Study Chair — Babylon University/ Iraq
Locations (1):
- Babylon University, Hillah, Babylon, Iraq

REFERENCES:
- [Derived] Hadwan MH, Almashhedy LA, Alsalman AR. Oral Zinc Supplementation Restores Superoxide Radical Scavengers to Normal Levels in Spermatozoa of Iraqi Asthenospermic Patients. Int J Vitam Nutr Res. 2015;85(3-4):165-73. doi: 10.1024/0300-9831/a000235. PMID 26780395